CLINICAL TRIAL: NCT05516758
Title: A Phase 2b, Double-Blind, Placebo-Controlled Study to Evaluate Peresolimab in Adult Participants With Moderately-to-Severely Active Rheumatoid Arthritis
Brief Title: A Study of Peresolimab (LY3462817) in Participants With Moderately-to-Severely Active Rheumatoid Arthritis
Acronym: RESOLUTION-1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to an unfavourable benefit-risk profile observed in interim data analysis.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18525; J1A-MC-KDAF (Other: Eli Lilly and Company); 2022-501425-20-00 (Other: EU Trial Number); U1111-1283-9566 (Other: Universal Trial Number)
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Results first posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Rheumatoid Arthritis; Arthritis; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases; Connective Tissue Diseases; Autoimmune Diseases; Immune System Diseases
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases; Connective Tissue Diseases; Autoimmune Diseases; Immune System Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Peresolimab 1000 mg SC Q4W (Experimental): Participants received peresolimab 1000 milligram (mg) subcutaneously (SC) once every 4 weeks (Q4W) from Week 0 to Week 24. At Week 24, based on their Clinical Disease Activity Index (CDAI) score, participants continued peresolimab 1000 mg SC Q4W from Week 24 to Week 60.
  Interventions: Drug: Peresolimab
- Peresolimab 1000 mg SC Q4W to Peresolimab 1000 mg SC Q12W (Experimental): Participants received peresolimab 1000 mg SC Q4W from Week 0 to Week 24. At Week 24, based on their CDAI score, participants switched to peresolimab 1000 mg SC once every 12 weeks (Q12W) from Week 24 to Week 60.
  Interventions: Drug: Peresolimab
- Peresolimab 400 mg SC Q4W (Experimental): Participants received peresolimab 400 mg SC Q4W from Week 0 to Week 24. At Week 24, based on their CDAI score, participants continued peresolimab 400 mg SC Q4W from Week 24 to Week 60.
  Interventions: Drug: Peresolimab
- Peresolimab 400 mg SC Q4W to Peresolimab 400 mg SC Q12W (Experimental): Participants received peresolimab 400 mg SC Q4W from Week 0 to Week 24. At Week 24, based on their CDAI score, participants switched to peresolimab 400 mg SC Q12W from Week 24 to Week 60.
  Interventions: Drug: Peresolimab
- Peresolimab 100 mg SC Q4W (Experimental): Participants received peresolimab 100 mg SC Q4W from Week 0 to Week 60.
  Interventions: Drug: Peresolimab
- Placebo SC Q4W to Peresolimab 1000 mg SC Q4W (Experimental): Participants received peresolimab-matched placebo SC Q4W from Week 0 to Week 12 and then switched to peresolimab 1000 mg SC Q4W from Week 12 to Week 60.
  Interventions: Drug: Peresolimab; Drug: Placebo
- Placebo SC Q4W to Peresolimab 400 mg SC Q4W (Experimental): Participants received peresolimab-matched placebo SC Q4W from Week 0 to Week 12 and then switched to peresolimab 400 mg SC Q4W from Week 12 to Week 60.
  Interventions: Drug: Peresolimab; Drug: Placebo

INTERVENTIONS:
Drug: Peresolimab — Administered SC
Drug: Placebo — Administered SC
  Arms: Placebo SC Q4W to Peresolimab 1000 mg SC Q4W; Placebo SC Q4W to Peresolimab 400 mg SC Q4W

SUMMARY:
The main purpose of this study is to assess the safety and efficacy of peresolimab in adult participants with moderately-to-severely active rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of adult onset rheumatoid arthritis (RA) for at least 3 months prior to screening, as defined by the 2010 ACR/European League Against Rheumatism (EULAR) classification criteria
* Have moderately-to-severely active RA, at screening and baseline, defined by the presence of

  * ≥6 swollen joints based on 66 joint count, and
  * ≥6 tender joints based on 68 joint count.
* Have had an inadequate response to, or loss of response or intolerance to at least 1 conventional synthetic DMARD (csDMARD), biologic DMARD ( bDMARD), or targeted synthetic DMARD (tsDMARD) treatment.

Exclusion Criteria:

* Have Class IV RA according to ACR revised criteria.
* Have presence of 1 or more significant concurrent medical conditions per investigator judgment, including but not limited to

  * poorly controlled diabetes or hypertension
  * chronic kidney disease stage IIIb, IV, or V
  * symptomatic heart failure according to New York Heart Association Class II, III, or IV
  * myocardial infarction, unstable angina pectoris, stroke or transient ischemic attack, within the past 12 months before randomization
  * severe chronic pulmonary disease, for example, requiring oxygen therapy
  * major chronic inflammatory disease or connective tissue disease other than RA, including but not limited to,

    * systemic lupus erythematosus
    * psoriatic arthritis
    * axial spondyloarthritis including ankylosing spondylitis and non-radiographic axial spondyloarthritis
    * reactive arthritis
    * gout
    * scleroderma
    * polymyositis
    * dermatomyositis
    * active fibromyalgia, or
    * multiple sclerosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 491 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2025-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (130):
- United States (53):
  - Accel Research Sites - Birmingham Clinical Research Unit, Birmingham, Alabama
  - Arizona Arthritis & Rheumatology Research PLLC, Gilbert, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC, Glendale, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC, Mesa, Arizona
  - Arizona Arthritis & Rheumatology Associates, PLLC, Phoenix, Arizona
  - Medvin Clinical Research - Metyas, Covina, California
  - St Joseph Heritage Healthcare, Fullerton, California
  - Newport Huntington Medical Group, Huntington Beach, California
  - Desert Medical Advances, Rancho Mirage, California
  - Dan La, MD Inc, Tujunga, California
  - Wolverine Clinical Trials, Tustin, California
  - Medvin Clinical Research - Su, Whittier, California
  - Denver Arthritis Clinic, Denver, Colorado
  - Tekton Research - Fort Collins - East Harmony Road, Fort Collins, Colorado
  - HARAC Research Corp, Avon Park, Florida
  - Encore Medical Research of Boynton Beach, Boynton Beach, Florida
  - Clinical Research of West Florida, Inc. (Clearwater), Clearwater, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Baycare Medical Group, St. Petersburg, Florida
  - West Broward Rheumatology Associates, Tamarac, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Baycare Medical Group, Tampa, Florida
  - Great Lakes Clinical Trials - Ravenswood, Chicago, Illinois
  - Hinsdale Orthopaedics - llinois Bone & Joint Institute, Hinsdale, Illinois
  - Accurate Clinical Research, Lake Charles, Louisiana
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - AA Medical Research Center, Grand Blanc, Michigan
  - Arthritis and Rheumatology Center of MI - Rochester Hills, Rochester Hills, Michigan
  - Clinvest Research LLC, Springfield, Missouri
  - Saint Louis Rheumatology, St Louis, Missouri
  - Arthritis & Osteoporosis Associates - Freehold, Freehold, New Jersey
  - Albuquerque Center for Rheumatology, Albuquerque, New Mexico
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Joseph S. and Diane H. Steinberg Ambulatory Care Center, Brooklyn, New York
  - DJL Clinical Research, PLLC, Charlotte, North Carolina
  - Cape Fear Arthritis Care, Leland, North Carolina
  - Paramount Medical Research & Consulting, LLC, Middleburg Heights, Ohio
  - Health Research of Oklahoma, Oklahoma City, Oklahoma
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Piedmont Arthritis Clinic, Greenville, South Carolina
  - Tekton Research, Inc, Austin, Texas
  - Accurate Clinical Management, Baytown, Texas
  - Metroplex Clinical Research Center, Dallas, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Accurate Clinical Management - Houston, Houston, Texas
  - Accurate Clinical Research, Houston, Texas
  - Laila A Hassan, MD, PA, Houston, Texas
  - DM Clinical Research - Tomball, Tomball, Texas
  - DM Clinical Research/Rheumatology Clinic of Houston, Tomball, Texas
  - Sound Clinical Research, LLC, Bothell, Washington
  - Arthritis Northwest, PLLC, Spokane, Washington
  - Rheumatology & Pulmonary Clinic, Beckley, West Virginia
- Argentina (11):
  - Organizacion Medica de Investigacion, CABA, Buenos Aires
  - Centro Privado de Medicina Familiar / Mindout Research, Ciudad Autónoma de Buenos Aire, Buenos Aires
  - CIPREC, Buenos Aires, Buenos Aires F.D.
  - APRILLUS Asistencia E Investigacion, CABA, Buenos Aires F.D.
  - Clinica Adventista Belgrano, CABA, Ciudad Autónoma de Buenos Aire
  - Centro de Investigaciones Reumatológicas, San Miguel de Tucumán, Tucumán Province
  - Centro de Investigaciones Médicas Tucuman, San Miguel de Tucumán, Tucumán Province
  - Fundación Respirar, Buenos Aires
  - Hospital Córdoba, Córdoba
  - Instituto Medico Strusberg, Córdoba
  - Centro Polivalente de Asistencia e Investigacion Clinica - CER San Juan, San Juan
- Canada (3):
  - Aggarwal and Associates Limited, Brampton, Ontario
  - Centre de Recherche Musculo-Squelettique, Trois-Rivières, Quebec
  - G.R.M.O. (Groupe de recherche en maladies osseuses) Inc., Québec
- China (9):
  - Afflilated Hospital of Bengbu Medical College, Bengbu, Anhui
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong
  - ShenZhen People's Hospital, Shenzhen, Guangdong
  - Tongji Hospital Tongji Medical,Science & Technology, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Jiangxi Pingxiang People's Hospital, Pingxiang, Jiangxi
  - Huashan Hospital Affiliated Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
- Greece (5):
  - General Hospital of Athens Hippokratio, Athens, Attikí
  - General Hospital of Athens Laiko, Athens, Attikí
  - Attikon General University Hospital, Chaïdári, Attikí
  - University General Hospital of Heraklion, Heraklion, Krítí
  - University Hospital of Alexandroupolis, Alexandroupoli, Évros
- Hungary (3):
  - Revita Clinic, Budapest, Pest County
  - Vital Medical Center, Veszprém, Veszprém City
  - Qualiclinic, Budapest
- Japan (21):
  - Chubu Rosai Hospital, Nagoya, Aichi-ken
  - Koujunkai Daido Clinic, Nagoya, Aichi-ken
  - Juntendo University Urayasu Hospital, Urayasu, Chiba
  - Shinkokura Hospital, Kitakyushu, Fukuoka
  - Tobata General Hospital, Kitakyushu, Fukuoka
  - University of Occupational and Enviromental Health, Kitakyushu, Fukuoka
  - Sagawa Akira Rheumatology Clinic, Sapporo, Hokkaido
  - Tonan Hospital, Sapporo, Hokkaido
  - Yoshida Internal Medicine Clinic, Sakaki, Nagano
  - Sasebo Chuo Hospital, Sasebo, Nagasaki
  - Nagaoka Red Cross Hospital, Nagaoka, Niigata
  - Hirose Clinic - Tokorozawa, Tokorozawa, Saitama
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - National Hospital Organization Chibahigashi National Hospital, Chiba
  - Hiroshima Clinic, Hiroshima
  - Hiroshima University Hospital, Hiroshima
  - Bayside Misato Medical Center, Kochi
  - Shinonoi General Hospital, Nagano
  - Nagasaki Internal Medicine- Rheumatology Hospital, Nagasaki
  - Okayama City General Medical Center Okayama City Hospital, Okayama
  - Machida Municipal Hospital, Tokyo
- Mexico (5):
  - Centro Medico del Angel, Mexicali, Estado de Baja California
  - Clinica de Investigacion en Reumatologia y Obesidad S. C., Guadalajara, Jalisco
  - Clinstile, S.A. de C.V., Mexico City, Mexico City
  - Kohler and Milstein Research S.A. de C.V., Mérida, Yucatán
  - Investigacion y Biomedicina de Chihuahua, Chihuahua City
- Poland (10):
  - Ai Centrum Medyczne Sp. Z O.O. Sp.K., Poznan, Greater Poland Voivodeship
  - Twoja Przychodnia Poznanskie Centrum Medyczne, Poznan, Greater Poland Voivodeship
  - Szpital Uniwersytecki Nr 2 w Bydgoszczy, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Twoja Przychodnia NCM, Nowa Sól, Lubusz Voivodeship
  - MICS Centrum Medyczne Warszawa, Warsaw, Masovian Voivodeship
  - Rheuma Medicus- Zak��ad Opieki Zdrowotnej, Warsaw, Masovian Voivodeship
  - Centrum Medyczne Reuma Park, Warsaw, Masovian Voivodeship
  - Nova Reuma Społka Partnerska, Bialystok, Podlaskie Voivodeship
  - Nzoz Bif-Med, Bytom, Silesian Voivodeship
  - Ambulatorium Sp. z o.o., Elblag, Warmian-Masurian Voivodeship
- Puerto Rico (4):
  - Centro Reumatologico Caguas, Caguas
  - Latin Clinical Trial Center, San Juan
  - GCM Medical Group, PSC - Hato Rey Site, San Juan
  - Mindful Medical Research, San Juan
- Spain (6):
  - CHUAC-Complejo Hospitalario Universitario A Coruña, A Coruña, A Coruña [La Coruña]
  - Clínica Gaias - Santiago, Santiago de Compostela, A Coruña [La Coruña]
  - Osi Bilbao-Basurto, Bilbao, Basque Country
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - CHUS - Hospital Clinico Universitario, Santiago de Compostela, Galicia [Galicia]
  - Hospital Quiron Infanta Luisa, Seville

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement
Supporting Information: Study Protocol, SAP, CSR
Time Frame: : Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A Study of Peresolimab (LY3462817) in Participants With Moderately-to-Severely Active Rheumatoid Arthritis (RESOLUTION-1) — https://trials.lilly.com/en-US/trial/356796

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Peresolimab 1000 mg SC Q4W | Peresolimab 1000 mg SC Q4W to Peresolimab 1000 mg SC Q12W | Peresolimab 400 mg SC Q4W | Peresolimab 400 mg SC Q4W to Peresolimab 400 mg SC Q12W | Peresolimab 100 mg SC Q4W | Placebo SC Q4W to Peresolimab 1000 mg SC Q4W | Placebo SC Q4W to Peresolimab 400 mg SC Q4W
Started | 115 | 26 | 116 | 25 | 69 | 73 | 67
Received Atleast One Dose of Study Drug | 115 | 26 | 116 | 25 | 68 | 73 | 67
Peresolimab 1000 mg Q4W (Discontinued Before Week 24) (Safety Analysis Population: All randomized participants who received at least one dose of study drug. Participants were analyzed based on the actual treatment they received throughout the study period.) | 12 | 0 | 0 | 0 | 0 | 0 | 0
Peresolimab 1000 mg Q4W to Peresolimab 1000 mg Q4W (Safety Analysis Population: Participants who received peresolimab 1000 mg SC Q4W throughout the study (Weeks 0-60).) | 103 | 0 | 0 | 0 | 0 | 0 | 0
Peresolimab 400 mg Q4W (Discontinued Before Week 24) (Safety Analysis Population: All randomized participants who received at least one dose of study drug. Participants were analyzed based on the actual treatment they received throughout the study period.) | 0 | 0 | 22 | 0 | 0 | 0 | 0
Peresolimab 400 mg Q4W to Peresolimab 400 mg Q4W (Safety Analysis Population: Participants who received peresolimab 400 mg SC Q4W throughout the study (Weeks 0-60).) | 0 | 0 | 94 | 0 | 0 | 0 | 0
Placebo SC Q4W Only (Safety Analysis Population: Placebo SC Q4W only = 14: Included 7 participants from the "Placebo to peresolimab 1000 mg Q4W" arm and 7 participants from the "Placebo to peresolimab 400 mg SC Q4W" arm who received placebo SC Q4W only and discontinued before Week 12. For analyses, based on the actual treatment received, these participants were analyzed together.) | 0 | 0 | 0 | 0 | 0 | 7 | 7
Placebo SC Q4W to Peresolimab 1000 mg SC Q4W (Safety Analysis Population: All randomized participants who received at least one dose of study drug. Participants were analyzed based on the actual treatment they received throughout the study period.) | 0 | 0 | 0 | 0 | 0 | 66 | 0
Placebo SC Q4W to Peresolimab 400 mg SC Q4W (Safety Analysis Population: All randomized participants who received at least one dose of study drug. Participants were analyzed based on the actual treatment they received throughout the study period.) | 0 | 0 | 0 | 0 | 0 | 0 | 60
Completed | 78 | 23 | 73 | 22 | 48 | 47 | 36
Not Completed | 37 | 3 | 43 | 3 | 21 | 26 | 31
Not completed — Adverse Event | 5 | 1 | 3 | 0 | 1 | 3 | 5
Not completed — Assigned treatment by mistake | 1 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 6 | 0 | 2 | 0 | 3 | 6 | 3
Not completed — Lost to Follow-up | 2 | 0 | 2 | 0 | 3 | 2 | 1
Not completed — Other- As reported by the site | 2 | 1 | 8 | 1 | 2 | 3 | 8
Not completed — Physician Decision | 1 | 0 | 7 | 0 | 1 | 1 | 2
Not completed — Protocol Deviation | 1 | 0 | 0 | 0 | 0 | 1 | 5
Not completed — Withdrawal by Subject | 11 | 1 | 15 | 2 | 7 | 7 | 6
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Non-compliance With Study Drug | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Site Terminated by Sponsor | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 4 | 0 | 3 | 0 | 2 | 3 | 0
Not completed — Participants not proceeding to Follow-up phase | 1 | 0 | 2 | 0 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug. As pre-specified in the statistical analysis plan (SAP), participants receiving the same initial treatment were grouped together based on treatment from Week 0 to Week 12 (Placebo) and Week 0 to Week 24 (Peresolimab 1000 mg and 400 mg groups).
Groups:
- Peresolimab 1000 mg SC Q4W: All participants who initially received peresolimab 1000 mg SC Q4W from Week 0 to Week 24 were grouped together and reported.
- Peresolimab 400 mg SC Q4W: All participants who initially received peresolimab 400 mg SC Q4W from Week 0 to Week 24 were grouped together and reported.
- Peresolimab 100 mg SC Q4W: All participants who received peresolimab 100 mg SC Q4W from Week 0 to Week 60 were reported.
- Placebo SC Q4W: All participants received peresolimab-matched Placebo SC Q4W from Week 0 to Week 12 were grouped together and reported.
- Total: Total of all reporting groups
Arm/Group | Peresolimab 1000 mg SC Q4W | Peresolimab 400 mg SC Q4W | Peresolimab 100 mg SC Q4W | Placebo SC Q4W | Total
Number analyzed (Participants) | 141 | 141 | 68 | 140 | 490
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.20 (11.73) | 54.50 (11.56) | 54.40 (12.08) | 54.00 (10.15) | 54.00 (11.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 119 | 52 | 114 | 404
  Male | 22 | 22 | 16 | 26 | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 72 | 73 | 44 | 78 | 267
  Not Hispanic or Latino | 67 | 67 | 24 | 57 | 215
  Unknown or Not Reported | 2 | 1 | 0 | 5 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 10 | 14 | 6 | 22 | 52
  Asian | 20 | 17 | 6 | 14 | 57
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 2 | 2 | 4 | 13
  White | 105 | 106 | 54 | 99 | 364
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 0 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 36 | 39 | 24 | 36 | 135
  Canada | 0 | 2 | 1 | 0 | 3
  China | 6 | 8 | 4 | 7 | 25
  Greece | 1 | 1 | 0 | 0 | 2
  Hungary | 11 | 6 | 2 | 10 | 29
  Japan | 14 | 9 | 2 | 7 | 32
  Mexico | 18 | 21 | 8 | 27 | 74
  Poland | 19 | 24 | 11 | 12 | 66
  Spain | 2 | 1 | 1 | 8 | 12
  United States | 34 | 30 | 15 | 33 | 112

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving 20% Improvement in American College of Rheumatology Criteria (ACR20) Response at Week 12
Description: The ACR20 response was a composite measure of clinical, laboratory, and functional assessments used to evaluate improvement in rheumatoid arthritis signs and symptoms. ACR20 responders were participants with at least 20% improvement from baseline in tender joint count (TJC) and swollen joint count (SJC), and at least 20% improvement in 3 of the 5 remaining core measures: Patient's Assessment of Arthritis Pain, Patient's Global Assessment of Disease Activity, Physician's Global Assessment of Disease Activity, Health Assessment Questionnaire-Disability Index (HAQ-DI) which measures participants' perceived degree of difficulty performing daily activities, and acute phase reactant as measured by high-sensitivity C-reactive protein (hsCRP). Percentage of participants achieving ACR20 response= (number of ACR20 responders)/ (number of participants analyzed) *100.
Time Frame: Week 12
Population: All randomized participants who received atleast one dose of study drug. Non-Responder Imputation (NRI) was applied for participants who had missing data, used rescue or prohibited medication or early discontinued from study or study intervention before or at Week 12. As pre-specified in the SAP, participants receiving the same initial treatment were grouped together based on treatment from Week 0 to Week 12 (Placebo) and Week 0 to Week 24 (Peresolimab 1000 mg and 400 mg groups).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Placebo SC Q4W: All participants received peresolimab -matched placebo SC Q4W from Week 0 to Week 12 were grouped together and reported.
Arm/Group | Peresolimab 1000 mg SC Q4W | Peresolimab 400 mg SC Q4W | Peresolimab 100 mg SC Q4W | Placebo SC Q4W
Number analyzed (Participants) | 141 | 141 | 68 | 140
Percentage of Participants | 51.8 [43.5 to 60.0] | 51.1 [42.8 to 59.3] | 44.1 [32.3 to 55.9] | 39.3 [31.2 to 47.4]
Statistical Analysis 1: Comparison: Peresolimab 1000 mg SC Q4W vs Placebo SC Q4W; Test type: Superiority; p = 0.014, Regression, Logistic; Odds Ratio (OR) = 1.88, 95% CI 2-sided [1.14 to 3.11]
Statistical Analysis 2: Comparison: Peresolimab 400 mg SC Q4W vs Placebo SC Q4W; Test type: Superiority; p = 0.098, Regression, Logistic; Odds Ratio (OR) = 1.53, 95% CI 2-sided [0.92 to 2.52]
Statistical Analysis 3: Comparison: Peresolimab 100 mg SC Q4W vs Placebo SC Q4W; Test type: Superiority; p = 0.534, Regression, Logistic; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.66 to 2.23]

2. Secondary Outcome: Percentage of Participants Achieving 50% Improvement in American College of Rheumatology Criteria (ACR50) Response at Week 12
Description: The ACR50 response was a composite measure of clinical, laboratory, and functional assessments used to evaluate improvement in rheumatoid arthritis signs and symptoms. ACR50 responders were participants with at least 50% improvement from baseline in TJC and SJC, and at least 50% improvement in 3 of the 5 remaining core measures: Patient's Assessment of Arthritis Pain, Patient's Global Assessment of Disease Activity, Physician's Global Assessment of Disease Activity, HAQ-DI which measures participants' perceived degree of difficulty performing daily activities, and acute phase reactant as measured by hsCRP. Percentage of participants achieving ACR50 response = (number of ACR50 responders) / (number of participants analyzed) * 100.
Time Frame: Week 12
Population: All randomized participants who received atleast one dose of study drug. NRI was applied for participants who had missing data, used rescue or prohibited medication or early discontinued from study or study intervention before or at Week 12. As pre-specified in the SAP, participants receiving the same initial treatment were grouped together based on treatment from Week 0 to Week 12 (Placebo) and Week 0 to Week 24 (Peresolimab 1000 mg and 400 mg groups).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Peresolimab 1000 mg SC Q4W | Peresolimab 400 mg SC Q4W | Peresolimab 100 mg SC Q4W | Placebo SC Q4W
Number analyzed (Participants) | 141 | 141 | 68 | 140
Percentage of Participants | 22.7 [15.8 to 29.6] | 19.1 [12.7 to 25.6] | 11.8 [4.1 to 19.4] | 10.7 [5.6 to 15.8]

3. Secondary Outcome: Percentage of Participants Achieving 70% Improvement in American College of Rheumatology Criteria (ACR70) Response at Week 12
Description: The ACR70 response was a composite measure of clinical, laboratory, and functional assessments used to evaluate improvement in rheumatoid arthritis signs and symptoms. ACR70 responders were participants with at least 70% improvement from baseline in TJC and SJC, and at least 70% improvement in 3 of the 5 remaining core measures: Patient's Assessment of Arthritis Pain, Patient's Global Assessment of Disease Activity, Physician's Global Assessment of Disease Activity, HAQ-DI which measures participants' perceived degree of difficulty performing daily activities, and acute phase reactant as measured by hsCRP. Percentage of participants achieving ACR70 response = (number of ACR70 responders) / (number of participants analyzed) * 100.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Peresolimab 1000 mg SC Q4W | Peresolimab 400 mg SC Q4W | Peresolimab 100 mg SC Q4W | Placebo SC Q4W
Number analyzed (Participants) | 141 | 141 | 68 | 140
Percentage of Participants | 7.1 [2.9 to 11.3] | 6.4 [2.3 to 10.4] | 7.4 [1.1 to 13.6] | 2.9 [0.1 to 5.6]

4. Secondary Outcome: Percentage of Participants With Low Disease Activity (LDA) According to Disease Activity Score Modified to Include the 28 Diarthrodial Joint Count-High-Sensitivity C-Reactive Protein (DAS28-hsCRP) ≤3.2 at Week 12
Description: DAS28-hsCRP LDA was defined as DAS28-hsCRP score of ≤3.2. The Disease Activity Score (DAS) based on 28 joint counts consisted of a composite numerical score derived from the following variables: tender joint count (0 to 28), swollen joint count (0 to 28), high-sensitivity C-reactive protein (hsCRP, mg/mL), and the patient's global assessment of disease activity. DAS28-hsCRP was calculated using following formula: DAS28-hsCRP equals to (=) 0.56*square root (sqrt) (TJC28) plus (+) 0.28*sqrt (SJC28)+ 0.014* participant's global assessment of disease activity+ 0.36*natural log(hsCRP+1) + 0.96. Total Scores ranged from 1.0 to 9.4, with lower scores indicating less disease activity.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Peresolimab 1000 mg SC Q4W | Peresolimab 400 mg SC Q4W | Peresolimab 100 mg SC Q4W | Placebo SC Q4W
Number analyzed (Participants) | 141 | 141 | 68 | 140
Percentage of Participants | 17.7 [11.4 to 24.0] | 17.0 [10.8 to 23.2] | 17.6 [8.6 to 26.7] | 7.1 [2.9 to 11.4]

5. Secondary Outcome: Percentage of Participants With Remission According to DAS28-hsCRP Score <2.6 at Week 12
Description: DAS28-hsCRP remission is defined as DAS28-hsCRP <2.6. DAS based on 28 joints consisted of composite numerical score of the following variables: tender joint count (TJC28), swollen joint count (SJC28), hsCRP (mg/mL), and patient's global assessment of disease activity. DAS28-hsCRP was calculated using following formula: DAS28-hsCRP=0.56*sqrt (TJC28) + 0.28*sqrt (SJC28) + 0.014* patient's global assessment of disease activity + 0.36*natural log(hsCRP+1) +0.96. Total Scores ranged from 1.0-9.4, where lower scores indicated less disease activity.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Peresolimab 1000 mg SC Q4W | Peresolimab 400 mg SC Q4W | Peresolimab 100 mg SC Q4W | Placebo SC Q4W
Number analyzed (Participants) | 141 | 141 | 68 | 140
Percentage of Participants | 11.3 [6.1 to 16.6] | 9.9 [5.0 to 14.9] | 5.9 [0.3 to 11.5] | 4.3 [0.9 to 7.6]

6. Secondary Outcome: Percentage of Participants Achieving LDA According to Clinical Disease Activity Index (CDAI) Score ≤10 at Week 12
Description: Low disease activity was defined as a CDAI score of ≤10. CDAI is a tool for measurement of disease activity in rheumatoid arthritis that does not require a laboratory component and was scored by the investigative site. It integrates TJC28 (scored 0-28 with higher scores indicating higher disease activity), SJC28 (scored 0-28 with higher scores indicating higher disease activity), Patient's Global Assessment of Disease Activity (scored on a visual analogue scale from 0-10 cm with higher scores indicating higher disease activity), and Physician's Global Assessment of Disease Activity (scored on a visual analogue scale from 0-10 cm with higher scores indicating higher disease activity). CDAI is calculated by summing the values of the 4 components. CDAI scores range from 0 to 76; lower scores indicated lower disease activity.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Peresolimab 1000 mg SC Q4W | Peresolimab 400 mg SC Q4W | Peresolimab 100 mg SC Q4W | Placebo SC Q4W
Number analyzed (Participants) | 141 | 141 | 68 | 140
Percentage of Participants | 22.7 [15.8 to 29.6] | 20.6 [13.9 to 27.2] | 17.6 [8.6 to 26.7] | 12.1 [6.7 to 17.6]

7. Secondary Outcome: Percentage of Participants Achieving Remission According to CDAI Score ≤2.8 at Week 12
Description: Remission was defined as a CDAI score of ≤2.8. CDAI is a tool for measurement of disease activity in rheumatoid arthritis that does not require a laboratory component and was scored by the investigative site. It integrates TJC28 (scored 0-28 with higher scores indicating higher disease activity), SJC28 (scored 0-28 with higher scores indicating higher disease activity), Patient's Global Assessment of Disease Activity (scored on a visual analogue scale from 0-10 cm with higher scores indicating higher disease activity), and Physician's Global Assessment of Disease Activity (scored on a visual analogue scale from 0-10 cm with higher scores indicating higher disease activity). The CDAI is calculated by summing the values of the 4 components. CDAI scores range from 0 to 76; lower scores indicated lower disease activity.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Peresolimab 1000 mg SC Q4W | Peresolimab 400 mg SC Q4W | Peresolimab 100 mg SC Q4W | Placebo SC Q4W
Number analyzed (Participants) | 141 | 141 | 68 | 140
Percentage of Participants | 2.8 [0.1 to 5.6] | 5.7 [1.9 to 9.5] | 1.5 [0.0 to 4.3] | 1.4 [0.0 to 3.4]

8. Secondary Outcome: Change From Baseline in DAS28-hsCRP Score at Week 12
Description: DAS based on 28 joints consisted of composite numerical score of the following variables: tender joint count (TJC28), swollen joint count (SJC28), hsCRP (mg/mL), and patient's global assessment of disease activity. DAS28-hsCRP was calculated using following formula: DAS28-hsCRP = 0.56*sqrt (TJC28) + 0.28*sqrt (SJC28)+ 0.014* patient's global assessment of disease activity + 0.36*natural log(hsCRP+1) +0.96. Total scores ranged 1.0-9.4; lower scores indicated lower disease activity. A negative change from baseline indicates improvement in condition. Least Square (LS) Mean was calculated using mixed model repeated measures (MMRM) with treatment, stratification factors, baseline value, visit, treatment-by-visit interaction as fixed factors and participant as a random factor.
Time Frame: Baseline, Week 12
Population: All randomized participants who received atleast one dose of study drug and had data for DAS28-hsCRP. As pre-specified in the SAP, participants receiving the same initial treatment were grouped together based on treatment from Week 0 to Week 12 (Placebo) and Week 0 to Week 24 (Peresolimab 1000 mg and 400 mg groups).
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Peresolimab 1000 mg SC Q4W | Peresolimab 400 mg SC Q4W | Peresolimab 100 mg SC Q4W | Placebo SC Q4W
Number analyzed (Participants) | 133 | 123 | 66 | 126
Units on a scale | -1.67 [-1.89 to -1.46] | -1.41 [-1.63 to -1.19] | -1.29 [-1.59 to -0.99] | -1.08 [-1.30 to -0.85]

9. Secondary Outcome: Change From Baseline in CDAI Score at Week 12
Description: CDAI is a tool for measurement of disease activity in rheumatoid arthritis that does not require laboratory component and was scored by the investigative site. It integrates TJC28 (scored 0-28 with higher scores indicating higher disease activity), SJC28 (scored 0-28 with higher scores indicating higher disease activity), Patient's Global Assessment of Disease Activity (scored on a visual analogue scale from 0-10 cm with higher scores indicating higher disease activity), and Physician's Global Assessment of Disease Activity(scored on a visual analogue scale from 0-10 cm with higher scores indicating higher disease activity).CDAI is calculated by summing values of 4 components. CDAI scores range from 0 to 76; lower scores indicated lower disease activity. Negative change from baseline indicates improvement. LS Mean was calculated using MMRM with treatment, stratification factors, baseline value, visit, treatment-by-visit interaction as fixed factors and participant as a random factor.
Time Frame: Baseline, Week 12
Population: All randomized participants who received atleast one dose of study drug and had data for CDAI. As pre-specified in the SAP, participants receiving the same initial treatment were grouped together based on treatment from Week 0 to Week 12 (Placebo) and Week 0 to Week 24 (Peresolimab 1000 mg and 400 mg groups).
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Peresolimab 1000 mg SC Q4W | Peresolimab 400 mg SC Q4W | Peresolimab 100 mg SC Q4W | Placebo SC Q4W
Number analyzed (Participants) | 131 | 123 | 65 | 125
units on a scale | -19.98 [-22.34 to -17.63] | -17.20 [-19.64 to -14.77] | -15.42 [-18.63 to -12.21] | -14.04 [-16.48 to -11.60]

10. Secondary Outcome: Change From Baseline in HAQ-DI Score at Week 12
Description: HAQ-DI was a patient-reported questionnaire used in rheumatoid arthritis to assess physical function over the past week. It covered 8 domains of daily living activities: dressing and grooming, arising, eating, walking, hygiene, reach, grip, and other activities. Each activity category consists of 2 to 3 items. Each item is scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Any activity requiring assistance from another individual or the use of an assistive device adjusts to a minimum score of 2 to represent a more limited functional status. Total score was computed as the sum of domain scores and divided by the number of domains answered. The total score ranges from 0 to 3, with higher scores indicating greater physical limitations. LS Mean was calculated using MMRM with treatment, stratification factors, baseline value, visit and treatment-by-visit interaction as fixed effects and participant as a random effect.
Time Frame: Baseline, Week 12
Population: All randomized participants who received atleast one dose of study drug and had data for HAQ-DI outcome. As pre-specified in the SAP, participants receiving the same initial treatment were grouped together based on treatment from Week 0 to Week 12 (Placebo) and Week 0 to Week 24 (Peresolimab 1000 mg and 400 mg groups).
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Peresolimab 1000 mg SC Q4W | Peresolimab 400 mg SC Q4W | Peresolimab 100 mg SC Q4W | Placebo SC Q4W
Number analyzed (Participants) | 135 | 131 | 67 | 127
units on a scale | -0.44 [-0.53 to -0.35] | -0.42 [-0.51 to -0.32] | -0.23 [-0.35 to -0.10] | -0.26 [-0.36 to -0.17]

11. Secondary Outcome: Minimum Observed Concentration of Peresolimab by Treatment-Emergent Anti-Drug Antibody (TE ADA) Status
Description: Minimum observed concentration of peresolimab was assessed and stratified by Treatment-Emergent Anti-Drug Antibody (TE-ADA) status (TE ADA positive and TE ADA negative).
  A TE ADA evaluable participant was defined as TE ADA positive if they met the following criteria:
  1. Had baseline status of ADA Not Present and at least 1 postbaseline status of ADA Present with titer ≥ 2×minimum required dilution (MRD) of the ADA assay (Treatment Induced TE ADA). The MRD of peresolimab is 1:10.
  2. Had baseline and postbaseline status of ADA Present, with the postbaseline titer being 2 dilutions (4-fold) greater than the baseline titer.
  TE-ADA negative participants were defined as those not meeting the TE ADA positive criteria.
Time Frame: Baseline through Week 12
Population: All randomized participants who received atleast one dose of study drug and had TE-ADA data for this outcome. Participants receiving the same initial treatment were grouped together based on treatment from Week 0 to Week 24 (Peresolimab 1000 mg and 400 mg groups). No study participant treated with peresolimab 1000 mg Q4W had a positive TE-ADA result up to Week 12; thus, zero participants analyzed and no data were collected.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Arm/Group | Peresolimab 1000 mg SC Q4W | Peresolimab 400 mg SC Q4W | Peresolimab 100 mg SC Q4W
Number analyzed (Participants) | 130 | 126 | 61
nanograms per milliliter
  TE-ADA Positive: number analyzed (Participants) | 0 | 2 | 4
  TE-ADA Positive |  | 2060 (28) | 487 (248)
  TE-ADA Negative: number analyzed (Participants) | 130 | 124 | 57
  TE-ADA Negative | 14700 (113) | 4800 (155) | 1150 (152)

ADVERSE EVENTS:
Time Frame: Baseline up to end of follow-up (up to 72 weeks)
Description: All randomized participants from the safety population. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Groups:
- Peresolimab 1000 mg SC Q4W (Discontinued Before Week 24): Participants who received peresolimab 1000 mg SC Q4W from Week 0 to Week 24 (discontinued before Week 24) were reported under this group.
- Peresolimab 1000 mg SC Q4W to Peresolimab 1000 mg SC Q4W: Participants who received peresolimab 1000 mg SC Q4W from Week 0 to Week 24, then continued peresolimab 1000 mg SC Q4W from Week 24 to Week 60 were reported under this group.
- Peresolimab 1000 mg SC Q4W to Peresolimab 1000 mg SC Q12W: Participants who received peresolimab 1000 mg SC Q4W from Week 0 to Week 24, then switched to peresolimab 1000 mg SC Q12W from Week 24 to Week 60 were reported under this group.
- Peresolimab 400 mg SC Q4W (Discontinued Before Week 24): Participants who received peresolimab 400 mg SC Q4W from Week 0 to Week 24 (discontinued before Week 24) were reported under this group.
- Peresolimab 400 mg SC Q4W to Peresolimab 400 mg SC Q4W: Participants who received peresolimab 400 mg SC Q4W from Week 0 to Week 24, then continued peresolimab 400 mg SC Q4W from Week 24 to Week 60 were reported under this group.
- Peresolimab 400 mg SC Q4W to Peresolimab 400 mg SC Q12W: Participants who received peresolimab 400 mg SC Q4W from Week 0 to Week 24, then switched to peresolimab 400 mg SC Q12W from Week 24 to Week 60 were reported under this group.
- Peresolimab 100 mg SC Q4W: Participants who received peresolimab 100 mg SC Q4W from Week 0 to Week 60 were reported under this group.
- Placebo SC Q4W Only: Participants who received peresolimab matched Placebo SC Q4W only from Week 0 to Week 12 were reported under this group.
- Placebo SC Q4W to Peresolimab 1000 mg SC Q4W: Participants who received peresolimab-matched Placebo SC Q4W from Week 0 to Week 12 and then switched to peresolimab 1000 mg SC Q4W from Week 12 to Week 60 were reported under this group.
- Placebo SC Q4W to Peresolimab 400 mg SC Q4W: Participants who received peresolimab-matched Placebo SC Q4W from Week 0 to Week 12 and then switched to peresolimab 400 mg SC Q4W from Week 12 to Week 60 were reported under this group.
Arm/Group | Peresolimab 1000 mg SC Q4W (Discontinued Before Week 24) | Peresolimab 1000 mg SC Q4W to Peresolimab 1000 mg SC Q4W | Peresolimab 1000 mg SC Q4W to Peresolimab 1000 mg SC Q12W | Peresolimab 400 mg SC Q4W (Discontinued Before Week 24) | Peresolimab 400 mg SC Q4W to Peresolimab 400 mg SC Q4W | Peresolimab 400 mg SC Q4W to Peresolimab 400 mg SC Q12W | Peresolimab 100 mg SC Q4W | Placebo SC Q4W Only | Placebo SC Q4W to Peresolimab 1000 mg SC Q4W | Placebo SC Q4W to Peresolimab 400 mg SC Q4W
All-Cause Mortality (participants affected / at risk) | 0/12 | 1/103 | 0/26 | 0/22 | 0/94 | 0/25 | 0/68 | 0/14 | 0/66 | 0/60
Serious Adverse Events (participants affected / at risk) | 3/12 | 11/103 | 1/26 | 3/22 | 8/94 | 3/25 | 4/68 | 4/14 | 7/66 | 6/60
Other Adverse Events (participants affected / at risk) | 6/12 | 70/103 | 16/26 | 9/22 | 60/94 | 13/25 | 48/68 | 9/14 | 40/66 | 29/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Peresolimab 1000 mg SC Q4W (Discontinued Before Week 24) (N=12) | Peresolimab 1000 mg SC Q4W to Peresolimab 1000 mg SC Q4W (N=103) | Peresolimab 1000 mg SC Q4W to Peresolimab 1000 mg SC Q12W (N=26) | Peresolimab 400 mg SC Q4W (Discontinued Before Week 24) (N=22) | Peresolimab 400 mg SC Q4W to Peresolimab 400 mg SC Q4W (N=94) | Peresolimab 400 mg SC Q4W to Peresolimab 400 mg SC Q12W (N=25) | Peresolimab 100 mg SC Q4W (N=68) | Placebo SC Q4W Only (N=14) | Placebo SC Q4W to Peresolimab 1000 mg SC Q4W (N=66) | Placebo SC Q4W to Peresolimab 400 mg SC Q4W (N=60)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Granuloma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dengue fever (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fracture displacement (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Splenic injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Elbow deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/8 (0) | 0/89 (0) | 0/22 (0) | 1/18 (1) | 0/79 (0) | 0/22 (0) | 0/52 (0) | 0 (0) | 0/56 (0) | 0/44 (0)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung adenocarcinoma stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/8 (0) | 0/89 (0) | 0/22 (0) | 0/18 (0) | 0/79 (0) | 1/22 (1) | 0/52 (0) | 0 (0) | 0/56 (0) | 0/44 (0)
Ovarian cancer stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/8 (0) | 1/89 (1) | 0/22 (0) | 0/18 (0) | 0/79 (0) | 0/22 (0) | 0/52 (0) | 0 (0) | 0/56 (0) | 0/44 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalitis autoimmune (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 0/8 (0) | 1/89 (1) | 0/22 (0) | 0/18 (0) | 0/79 (0) | 0/22 (0) | 0/52 (0) | 0 (0) | 0/56 (0) | 0/44 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Peresolimab 1000 mg SC Q4W (Discontinued Before Week 24) (N=12) | Peresolimab 1000 mg SC Q4W to Peresolimab 1000 mg SC Q4W (N=103) | Peresolimab 1000 mg SC Q4W to Peresolimab 1000 mg SC Q12W (N=26) | Peresolimab 400 mg SC Q4W (Discontinued Before Week 24) (N=22) | Peresolimab 400 mg SC Q4W to Peresolimab 400 mg SC Q4W (N=94) | Peresolimab 400 mg SC Q4W to Peresolimab 400 mg SC Q12W (N=25) | Peresolimab 100 mg SC Q4W (N=68) | Placebo SC Q4W Only (N=14) | Placebo SC Q4W to Peresolimab 1000 mg SC Q4W (N=66) | Placebo SC Q4W to Peresolimab 400 mg SC Q4W (N=60)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 6 (7) | 1 (1) | 0 (0) | 4 (5) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Atrial escape rhythm (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bundle branch block right (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiomegaly (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Left atrial enlargement (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial fibrosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ventricular hypokinesia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid mass (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Age-related macular degeneration (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Episcleritis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye discharge (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scleritis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ulcerative keratitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrophic glossitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 4 (5) | 0 (0) | 0 (0) | 1 (3)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epiploic appendagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip erosion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug intolerance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Dystrophic calcification (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibrosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Injection site papule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 6 (8) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (5) | 0 (0) | 1 (1) | 2 (4)
Injection site urticaria (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lithiasis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Necrosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Biliary dyspepsia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Metabolic dysfunction-associated liver disease (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mite allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess soft tissue (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acarodermatitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asymptomatic bacteriuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacterial vaginosis (Infections and infestations) | 0/8 (0) | 0/89 (0) | 0/22 (0) | 0/18 (0) | 0/79 (0) | 0/22 (0) | 0/52 (0) | 0 (0) | 0/56 (0) | 1/44 (1)
Bacterial vulvovaginitis (Infections and infestations) | 0/8 (0) | 1/89 (1) | 0/22 (0) | 0/18 (0) | 0/79 (0) | 0/22 (0) | 0/52 (0) | 0 (0) | 0/56 (0) | 0/44 (0)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 6 (6) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Bursitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervicitis (Infections and infestations) | 0/8 (0) | 1/89 (1) | 0/22 (0) | 0/18 (0) | 0/79 (0) | 0/22 (0) | 0/52 (0) | 0 (0) | 0/56 (0) | 0/44 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 1 (1) | 6 (6) | 1 (1) | 1 (1) | 6 (6) | 1 (1) | 1 (1) | 0 (0) | 6 (7) | 3 (3)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dengue fever (Infections and infestations) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Dermatitis infected (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Gastroenteritis astroviral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hepatic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 3 (3) | 0 (0) | 3 (3) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 6 (6) | 3 (8) | 1 (1) | 3 (3) | 1 (1) | 6 (7) | 0 (0) | 3 (3) | 2 (2)
Oral fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 4 (6) | 0 (0) | 0 (0) | 3 (6) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 2 (2)
Pharyngitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Trichomoniasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 7 (8) | 0 (0) | 0 (0) | 5 (8) | 0 (0) | 9 (11) | 1 (1) | 3 (9) | 5 (6)
Upper respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 10 (12) | 0 (0) | 0 (0) | 8 (10) | 2 (2) | 6 (7) | 1 (1) | 3 (3) | 3 (4)
Viral diarrhoea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0/8 (0) | 0/89 (0) | 0/22 (0) | 0/18 (0) | 1/79 (1) | 0/22 (0) | 0/52 (0) | 0 (0) | 0/56 (0) | 0/44 (0)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fracture displacement (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immunisation reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lipohaemarthrosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal column injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic ulcer (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid intima-media thickness increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheterisation cardiac (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram pr shortened (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram repolarisation abnormality (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram st segment abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram t wave abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary occult blood positive (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Food intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 2 (2)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Greater trochanteric pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenosis sclerosing (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blepharal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ependymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/8 (0) | 1/89 (1) | 0/22 (0) | 0/18 (0) | 0/79 (0) | 0/22 (0) | 0/52 (0) | 0 (0) | 1/56 (1) | 0/44 (0)
Bell's palsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 2 (3) | 4 (5)
Intercostal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Affective disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (3) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0/8 (0) | 0/89 (0) | 0/22 (0) | 0/18 (0) | 0/79 (0) | 0/22 (0) | 0/52 (0) | 0 (0) | 1/56 (1) | 0/44 (0)
Endometriosis (Reproductive system and breast disorders) | 0/8 (0) | 1/89 (1) | 0/22 (0) | 0/18 (0) | 0/79 (0) | 0/22 (0) | 0/52 (0) | 0 (0) | 0/56 (0) | 0/44 (0)
Genital haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0/8 (0) | 1/89 (1) | 0/22 (0) | 0/18 (0) | 0/79 (0) | 0/22 (0) | 0/52 (0) | 0 (0) | 0/56 (0) | 0/44 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0/8 (0) | 0/89 (0) | 0/22 (0) | 0/18 (0) | 0/79 (0) | 1/22 (1) | 0/52 (0) | 0 (0) | 0/56 (0) | 0/44 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0/8 (0) | 0/89 (0) | 0/22 (0) | 0/18 (0) | 0/79 (0) | 0/22 (0) | 1/52 (1) | 0 (0) | 0/56 (0) | 0/44 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Superficial inflammatory dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract operation (Surgical and medical procedures) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intra-uterine contraceptive device removal (Surgical and medical procedures) | 0/8 (0) | 0/89 (0) | 0/22 (0) | 0/18 (0) | 0/79 (0) | 0/22 (0) | 1/52 (1) | 0 (0) | 0/56 (0) | 0/44 (0)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Knee operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mass excision (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pacemaker generated rhythm (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Turbinectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine dilation and curettage (Surgical and medical procedures) | 0/8 (0) | 0/89 (0) | 0/22 (0) | 0/18 (0) | 1/79 (1) | 0/22 (0) | 0/52 (0) | 0 (0) | 0/56 (0) | 0/44 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 3 (3) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-05-31): https://cdn.clinicaltrials.gov/large-docs/58/NCT05516758/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-01): https://cdn.clinicaltrials.gov/large-docs/58/NCT05516758/SAP_001.pdf